CLINICAL TRIAL: NCT03618004
Title: Technique of Restriction of Blood Flow Associated With the Ergonomic Cycle of Upper Limbs in Women. A Randomized Pilot Study
Brief Title: Technique of Restriction of Blood Flow Associated With the Ergonomic Cycle of Upper Limbs in Women
Acronym: Kaatsu-BFR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Real Fundación Victoria Eugenia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Kaatsu-BFR
Record Dates: First submitted 2018-08-01; First posted 2018-08-07 (Actual); Last update posted 2018-11-27 (Actual); Status verified 2018-11

CONDITIONS: Women's Health: Female Athlete/Female Athlete Triad
Keywords: Restriction of blood flow; Anaerobic capacity; Subjective perception of effort; Wingate; Isometric strength
MeSH Terms: conditions — Female Athlete Triad Syndrome | interventions — Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): The intervention lasted 17 minutes each session, 2 weekly sessions were carried out, during 4 weeks. The training started with a warm-up on the hand bike without a load for 5 minutes. Later, we did a work of 3 series of 30 seconds, in maximum power, with 5 minutes of rest between them. The intensity was calculated by 0.048 kp.kg.
  The subjects of the experimental group made use of the restriction of blood flow, using a pressure cuff coupled in the most proximal region of the arm, 10 cm wide. The pressure was calculated based on the initial systolic pressure of the subjects.
  Interventions: Other: Experimental group
- Control group (Active Comparator): The intervention lasted 17 minutes each session, 2 weekly sessions were carried out, during 4 weeks. The training started with a warm-up on the hand bike without a load for 5 minutes. Later, we did a work of 3 series of 30 seconds, in maximum power, with 5 minutes of rest between them. The intensity was calculated by 0.048 kp.kg.
  The subjects in the control group did not use pressure cuffs.
  Interventions: Other: Control group

INTERVENTIONS:
Other: Experimental group — The intervention lasted 17 minutes each session, 2 weekly sessions were carried out, during 4 weeks. The training started with a warm-up on the hand bike without a load for 5 minutes. Later, we did a work of 3 series of 30 seconds, in maximum power, with 5 minutes of rest between them. The intensity was calculated by 0.048 kp.kg.
  The subjects of the experimental group made use of the restriction of blood flow, using a pressure cuff coupled in the most proximal region of the arm, 10 cm wide. The pressure was calculated based on the initial systolic pressure of the subjects.
  Arms: Experimental group
Other: Control group — The intervention lasted 17 minutes each session, 2 weekly sessions were carried out, during 4 weeks. The training started with a warm-up on the hand bike without a load for 5 minutes. Later, we did a work of 3 series of 30 seconds, in maximum power, with 5 minutes of rest between them. The intensity was calculated by 0.048 kp.kg.
  The subjects in the control group did not use pressure cuffs.
  Arms: Control group

SUMMARY:
Finding alternatives to improve variables such as strength and anaerobic resistance is a subject of highly studied clinical intervention. The use of vascular occlusion associated with physical exercise has shown efficacy in improving these aspects.

The objective is to analyze the effectiveness of upper limb training with vascular occlusion (Kaatsu training) for the improvement of isometric strength and anaerobic capacity in women aged 18 to 38 years.

Study design. Randomized, prospective, single-blind, follow-up clinical study. The selected sample will be randomized into two groups: experimental and control. The intervention will consist of ergonomic exercises with and without vascular occlusion. Isometric strength will be assessed with a manual dynamometer, anaerobic capacity and peak power (anaerobic alactic system) and average power (anaerobic lactic system) with the wingate test, and subjective perception of effort with the Borg scale. The intervention will last 4 weeks, with 3 weekly sessions of 10 minutes each. A descriptive statistical analysis will be carried out among the dependent and independent variables of both groups. With the Kolmogórov distribution normality test and with the Anova and t-student tests for analysis of repeated measures.

Expected results. The investigators intend to observe improvement of isometric biceps and triceps strength and the anaerobic capacity of the group treated with vascular occlusion.

DETAILED DESCRIPTION:
The use of peripheral vascular occlusion in low intensity resistance exercises is a simple, safe and effective method, indicated for healthy individuals or with cardio-respiratory diseases, in the prevention of atrophy due to disuse, within the post rehabilitation approach. -surgical intervention and to improve the performance of athletes. Several studies evaluated the use of blood flow restriction prior to aerobic and anaerobic exercises, with heterogeneous results, without consensus. With this, our research proposal is a pioneer, as there is no other study that has investigated the use of upper limb vascular occlusion during anaerobic activity in an arm ergometer cycle. This could benefit individuals who need to maintain their anaerobic conditioning and who, for some reason, are unable to use the lower limbs. In addition, it could benefit in the performance and improvement of the physical fitness of athletes in wheelchairs of various modalities, which have their functions preserved in the upper limbs. Only a similar study showed the efficacy of this intervention model, but in lower limbs. The prevalence of men in published studies of anaerobic capacity with the WinGate test, with few studies recruiting women, indicates the need to perform the study with a female sample.

ELIGIBILITY:
Inclusion Criteria:

* Women
* Between 18 and 40 years old
* Physically active
* Without orthopedic injuries that prevented them from carrying out the exercise protocol

Exclusion Criteria:

* Diagnosis of chronic musculoskeletal, neurological or cardiorespiratory diseases
* With diagnosis of arterial hypertension, deep vein thrombosis or diabetes
* Pregnant
* Not sign the informed consent document

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2018-04-12 (Actual); Study Completion 2018-08-02 (Actual)

PRIMARY OUTCOMES:
Change from baseline isometric strength of biceps after treatment and at 1 month | Screening visit, within the first seven days after treatment and after one month follow-up visit]
  A Lafayette Manual Muscle Testing System force dynamometer (model 01165, USA) was used. The subject was standing with the trunk straight, the shoulders in neutral position with the arms aligned to the trunk and the elbows in 90 degrees of flexion. The evaluator requested a maximum voluntary isometric muscle contraction in elbow flexion, maintaining it for 5 seconds. Three repetitions were performed, with 5 minutes of rest between each series, the reference value being the average of the value obtained between the 3 repetitions.

SECONDARY OUTCOMES:
Change from baseline isometric strength of triceps after treatment and at 1 month | Screening visit, within the first seven days after treatment and after one month follow-up visit
  A Lafayette Manual Muscle Testing System force dynamometer (model 01165, USA) was used. The subject was standing with the trunk straight, the shoulders in neutral position with the arms aligned to the trunk and the elbows in 90 degrees of flexion. The evaluator requested a maximum voluntary isometric muscle contraction in elbow extension, maintaining it for 5 seconds. Three repetitions were performed, with 5 minutes of rest between each series, the reference value being the average of the value obtained between the 3 repetitions.
Change from baseline peak power after treatment and at 1 month | Screening visit, within the first seven days after treatment and after one month follow-up visit
  The WinGate test was used. The equipment used was an ergonomic clico for upper limbs (Excite® top seat, technogyn, Brazil). Each subject was placed seated, so that the center of the glenohumeral joint was aligned with the axis of the cranks of the equipment, with 90 degrees of knee flexion, which were aligned with shoulders and feet. The horizontal distance was adjusted so that the elbows were not in maximum extension and allowing the comfort of the participants.
Change from baseline relative power peak after treatment and at 1 month | Screening visit, within the first seven days after treatment and after one month follow-up visit
  The WinGate test was used. The equipment used was an ergonomic clico for upper limbs (Excite® top seat, technogyn, Brazil). Each subject was placed seated, so that the center of the glenohumeral joint was aligned with the axis of the cranks of the equipment, with 90 degrees of knee flexion, which were aligned with shoulders and feet. The horizontal distance was adjusted so that the elbows were not in maximum extension and allowing the comfort of the participants.
Change from baseline medium power after treatment and at 1 month | Screening visit, within the first seven days after treatment and after one month follow-up visit
  The WinGate test was used. The equipment used was an ergonomic clico for upper limbs (Excite® top seat, technogyn, Brazil). Each subject was placed seated, so that the center of the glenohumeral joint was aligned with the axis of the cranks of the equipment, with 90 degrees of knee flexion, which were aligned with shoulders and feet. The horizontal distance was adjusted so that the elbows were not in maximum extension and allowing the comfort of the participants.
Change from baseline relative medium power after treatment and at 1 month | Screening visit, within the first seven days after treatment and after one month follow-up visit
  The WinGate test was used. The equipment used was an ergonomic clico for upper limbs (Excite® top seat, technogyn, Brazil). Each subject was placed seated, so that the center of the glenohumeral joint was aligned with the axis of the cranks of the equipment, with 90 degrees of knee flexion, which were aligned with shoulders and feet. The horizontal distance was adjusted so that the elbows were not in maximum extension and allowing the comfort of the participants.
Change from baseline fatigue index after treatment and at 1 month | Screening visit, within the first seven days after treatment and after one month follow-up visit
  The WinGate test was used. The equipment used was an ergonomic clico for upper limbs (Excite® top seat, technogyn, Brazil). Each subject was placed seated, so that the center of the glenohumeral joint was aligned with the axis of the cranks of the equipment, with 90 degrees of knee flexion, which were aligned with shoulders and feet. The horizontal distance was adjusted so that the elbows were not in maximum extension and allowing the comfort of the participants.
Change from baseline subjective perception of effort after treatment and at 1 month | Screening visit, within the first seven days after treatment and after one month follow-up visit
  The subjective perception of effort was evaluated with the Borg CR-10 scale. One minute after the end of the evaluation, the effort perceived by the subjects was quantified from 0 to 10, with 0 the minimum perceived effort and 10 the maximum.
Change from baseline heart rate after treatment and at 1 month | Screening visit, within the first seven days after treatment and after one month follow-up visit
  The heart rate was assessed through a cardiac frequency meter (model Onrhythm 310, Geonaute, France). The resting heart rates were evaluated and one minute after the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Rubén Cuesta-Barriuso, PhD, Principal Investigator — Universidad Europea de Madrid
Locations (1):
- Royal Victoria Eugenia Foundation, Madrid, Madird, Spain

IPD SHARING:
Plan to Share IPD: No